CLINICAL TRIAL: NCT00878228
Title: Antiemetic Prophylaxis for Postdischarge Nausea and Vomiting After Hip Arthroscopy
Acronym: PDNV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29015
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): The study group will receive intraoperative IV ondansetron and also postoperative oral ondansetron tablets (8 mg each day for two days).
  Interventions: Drug: Ondansetron
- Control Group (Placebo Comparator): The control group will receive IV ondansetron intraoperatively and then oral placebo tablets (for 2 days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ondansetron — The study group will receive 4 mg of IV ondansetron perioperatively and also postoperative oral ondansetron tablets (8 mg each day for two days). The tablets will be concealed in generic capsules prepared by the pharmacy at the Hospital for Special Surgery to make the ondansetron tablets indistinguishable from the placebos.
  Other Names: Zofran
  Arms: Study Group
Drug: Placebo — The control group will receive IV ondansetron intraoperatively and then oral placebo tablets (for 2 days). These placebo tablets will contain lactose and be indistinguishable from the study medication.
  Arms: Control Group

SUMMARY:
The study is a randomized placebo controlled trial to determine whether repeated postoperative prophylactic ondansetron ("Zofran") administration will prevent postoperative and/or postdischarge nausea and vomiting in patients undergoing ambulatory hip arthroscopy. Ondansetron will be administered in the intra- and post-operative period. These individuals will be followed on postoperative days 1, 2, and 3. It is hypothesized that the incidence of postdischarge nausea and vomiting (PDNV) will be significantly decreased by postoperative prophylactic administration of multiple doses of ondansetron (Zofran).

ELIGIBILITY:
Inclusion Criteria:

* All patients of Dr. Coleman or Dr. Kelly ages 18 to 65 undergoing arthroscopic hip surgery
* Planned use of neuraxial anesthesia
* Ability to follow study protocol
* Willing to complete daily diary and be interviewed daily for three days after discharge

Exclusion Criteria:

* Patients younger than 18 years old and older than 65
* Patients unable to undergo a spinal or epidural anesthetic
* Having nausea or vomiting within 24 hours of the surgery
* Receiving drugs with anti-emetic properties within 24 hours of the surgery (e.g Zofran, Compazine, Phenergan, Reglan)
* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months)
* Hypersensitivity and/or allergy to ondansetron
* Intraoperative use of any volatile anesthetic
* Contraindication to a short course of NSAIDs (renal failure, intolerance)
* Allergy or intolerance to Vicodin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques YaDeau, MD, PhD, Principal Investigator — Hosptial for Special Surgery
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Osoba D, Zee B, Warr D, Latreille J, Kaizer L, Pater J. Effect of postchemotherapy nausea and vomiting on health-related quality of life. The Quality of Life and Symptom Control Committees of the National Cancer Institute of Canada Clinical Trials Group. Support Care Cancer. 1997 Jul;5(4):307-13. doi: 10.1007/s005200050078. PMID 9257427
- [Background] Pan PH, Lee SC, Harris LC. Antiemetic prophylaxis for postdischarge nausea and vomiting and impact on functional quality of living during recovery in patients with high emetic risks: a prospective, randomized, double-blind comparison of two prophylactic antiemetic regimens. Anesth Analg. 2008 Aug;107(2):429-38. doi: 10.1213/ane.0b013e318172f992. PMID 18633020
- [Background] Gan TJ, Meyer TA, Apfel CC, Chung F, Davis PJ, Habib AS, Hooper VD, Kovac AL, Kranke P, Myles P, Philip BK, Samsa G, Sessler DI, Temo J, Tramer MR, Vander Kolk C, Watcha M; Society for Ambulatory Anesthesia. Society for Ambulatory Anesthesia guidelines for the management of postoperative nausea and vomiting. Anesth Analg. 2007 Dec;105(6):1615-28, table of contents. doi: 10.1213/01.ane.0000295230.55439.f4. PMID 18042859
- [Background] Apfel CC, Korttila K, Abdalla M, Kerger H, Turan A, Vedder I, Zernak C, Danner K, Jokela R, Pocock SJ, Trenkler S, Kredel M, Biedler A, Sessler DI, Roewer N; IMPACT Investigators. A factorial trial of six interventions for the prevention of postoperative nausea and vomiting. N Engl J Med. 2004 Jun 10;350(24):2441-51. doi: 10.1056/NEJMoa032196. PMID 15190136
- [Background] White PF, O'Hara JF, Roberson CR, Wender RH, Candiotti KA; POST-OP Study Group. The impact of current antiemetic practices on patient outcomes: a prospective study on high-risk patients. Anesth Analg. 2008 Aug;107(2):452-8. doi: 10.1213/ane.0b013e31817b842c. PMID 18633023
- [Background] White PF, Sacan O, Nuangchamnong N, Sun T, Eng MR. The relationship between patient risk factors and early versus late postoperative emetic symptoms. Anesth Analg. 2008 Aug;107(2):459-63. doi: 10.1213/ane.0b013e31817aa6e4. PMID 18633024
- [Background] Pavlin DJ, Chen C, Penaloza DA, Polissar NL, Buckley FP. Pain as a factor complicating recovery and discharge after ambulatory surgery. Anesth Analg. 2002 Sep;95(3):627-34, table of contents. doi: 10.1097/00000539-200209000-00025. PMID 12198050
- See also: This is the link to the Hospital for Special Surgery home website. — http://www.hss.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: The study group received intraoperative IV ondansetron and also postoperative oral ondansetron tablets (8 mg each day for two days).
- Control Group: The control group received IV ondansetron intraoperatively and then oral placebo tablets (for 2 days).
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 49 | 49
Completed | 39 | 37
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 39 | 37 | 76
Age Continuous [Mean (Standard Deviation); unit: years] — 98 patients were enrolled in the study, but 22 were excluded for various reasons. The remaining 76 patients were analyzed for the study.
  years | 42 (14) | 37 (11) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — 98 patients were enrolled in the study, but 22 were excluded for various reasons. The remaining 76 patients were analyzed for the study.
  Participants
    Female | 18 | 19 | 37
    Male | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea
Description: Percentage of participants with nausea
Time Frame: Postdischarge Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 39 | 37
percentage of participants | 46 | 54

2. Secondary Outcome: Severity of Nausea
Description: Percentage of participants reporting moderate or severe nausea in the first 24 hours
Time Frame: Postdischarge Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 39 | 37
percentage of participants | 23 | 32

3. Secondary Outcome: Impact of Nausea and Vomiting on Quality of Life
Description: Percentage of participants whose quality of life was impacted by nausea and vomiting
Time Frame: Postdischarge Day 1
Measure: Number; unit: percentage of participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 39 | 37
percentage of participants | 18 | 30

ADVERSE EVENTS:
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes